CLINICAL TRIAL: NCT00511121
Title: An Exploratory Phase II Study of the Combination of a Tyrosine Kinase Inhibitor (STI571) and a Pegylated Human Recombinant Interferon alfa2b (PEGINTRON) in the Treatment of Chronic Myeloid Leukemia in Chronic Phase
Brief Title: Study of the Combination of a Tyrosine Kinase Inhibitor (STI571) and a Pegylated Human Recombinant Interferon alfa2b (PEGINTRON)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bologna (Other)
Collaborators: Novartis (Industry); Schering-Plough (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CML 011
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2007-08-03 (Estimated); Status verified 2007-08

CONDITIONS: Chronic Myeloid Leukemia
Keywords: chronic myeloid leukemia; tyrosine kinase
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: STI571 and PEG INTRON

SUMMARY:
This is a phase II multicenter, open-label study designed to investigate the feasibility (tolerance, compliance and safety) of a combination of the tyrosine kinase inhibitor STI 571 (GLIVEC, Novartis Pharma) with a pegylated *-Interferon 2b (PEG INTRON). The rationale for testing this combination is that 1) aIFN is curently the first line agent for the treatment of CML, 2) the pegylated formulation of aIFN is more convenient and is better tolerated than the conventional formulation, 3) STI571 is currently the most promising investigational agent for the treatment of CML because it is targeted to the molecular bases of the disease, is effective also in the advanced phases of the disease, and is effective also in the cases who are resistant to aIFN, 4) the mechanisms of action of the two agents are different. Therefore the combination of STI571 and PEGINTRON is likely to provide the best treatment of CML and to be tested very soon in randomized phase III studies of efficacy. So far STI571 and PEGINTRON have been investigated separately. The present study is an exploratory study that has been planned with the aim of evaluating the adverse events and the safety of the combination, so as to identify a safe and tolerable regime that can be tested prospectively for efficacy in a subsequent, randomized phase III study. Based on available knowledge and data, STI571 is more specific and can be more effective than PEGINTRON. Therefore in this exploratory study STI571 is given a priority over PEGINTRON as to dose and dose adaptation. Sixty subjects with chronic phase CML, previously untreated with any one of study drugs, will be enrolled over a 3 months period and will be treated and studied for 12 months. The patients can be pretreated with hydroxyurea , whenever required, hence are treated with STI 571 at a fixed dose (400mg) and with PEG-Intron at doses ranging from 50 to 150 *g weekly (the first cohort of 20 patients at 50 *g/w, the second cohort of 20 patients at 100 *g/w and the third cohort of 20 patients at 150 *g/w). The response (hematologic, cytogenetic and molecular) to the combination treatment will be evaluated every 3 months, and the pharmacokinetics of study drugs will be studied in a sample of study patients. The duration of the study is 12 months, for a total trial time of 15 months.

DETAILED DESCRIPTION:
STI 571 and *IFN are the two single most effective agents for the treatment of CML. Their mechanisms of actions are different. Their toxicity is also different, but both spare normal hemopoietic stem cells. STI 571 is well tolerated, while conventional *IFN is poorly tolerated, especially in the elderly. PEG *IFNs are going to substitute for conventional *IFNs because of a better pharmacokinetic and toxicity profile and because require less injections (once a week vs. once a day).Resistance to IFN (6-13) and to STI571 (29-34) occurs in vitro and in vivo, where it increases with time for IFN and is also expected to increase with time for STI571. STI571 and IFN have different mechanisms of action and it has been shown in vitro that the combination of STI571 with alfaIFN is more toxic than either agent alone against Ph positive cells (35-37). Therefore, a combination of STI 571 with a PEG *IFN is worth testing. A phase II, dose-finding, exploratory study is required to investigate feasibility, toxicity, safety and tolerability of the combination. In CML, PEG INTRON studies are more advanced than PEGASIS studies. These considerations provide the rationale for this phase II study of STI 571 and PEG INTRON in CML.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. First chronic phase
3. Performance status (ECOG/WHO) < or = 2
4. Written informed consent

Exclusion Criteria:

1. Age <18 or >65 years
2. Second chronic, accelerated or blastic phase
3. Performance status (ECOG/WHO) > 2
4. Inability to provide written informed consent
5. Prior treatment with STI 571 or alfaIFN
6. Prior alloBMT
7. Prior autoBMT
8. Prior non-conventional, intensive chemotherapy in the last 12 months
9. Prior experimental agents in the last 60 days
10. Prior conventional chemotherapy in the last 60 days (in case of Busulfan or other alkylating agents) or in the last 10 days (in case of Hydroxyurea or other cell-cycle dependent drugs)
11. Pregnancy
12. Formal refusal of any recommendation of a safe contraception
13. Alcohol or drug addiction
14. Positivity for HBV, HCV or HIV
15. Altered hepatic or renal function as defined by AST/ALT or bilirubine > 3 times upper normal limits (UNL) and by creatinine > or = 20mg/L
16. Any other disease or condition that by the advise of the responsible physician would make the treatment dangerous for the patient or would make the patient ineligible for the study, including physical, psychiatric, social and behavioural problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5
Dates: Start 2001-04

PRIMARY OUTCOMES:
This is a study that is designed to determine the AE and the safety of a combination of standard dose of STI 571 (400 my daily) with a low-intermediate dose of *IFN (50 t0 150 ug weekly) and the compliane of the patients to the combination.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Baccarani, MD, Principal Investigator — Istituto di Ematologia "L e A Seragnoli" Bologna